CLINICAL TRIAL: NCT02576600
Title: Pupillometry Guided Versus Standard Practice Remifentanil Administration and Total Opioid Consumption
Brief Title: Pupillometry Guided Remifentanil Administration and Total Opioid Consumption During Propofol - Remifentanil TCI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pr Isabelle CONSTANT (Other)
Responsible Party: Sponsor-Investigator, Pr Isabelle CONSTANT, Professor Isabelle Constant, Hôpital Armand Trousseau
Organization: Hôpital Armand Trousseau (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Anesthesie Trousseau 001
Record Dates: First submitted 2015-10-13; First posted 2015-10-15 (Estimated); Last update posted 2015-10-19 (Estimated); Status verified 2015-10

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Propofol; Remifentanil

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PUPILLO (Experimental): Videopupillometer Algiscan peroperative remifentanil target concentration adapted every five minutes to pupillary diameter in patients under propofol and remifentanil TCI
  Interventions: Device: Videopupillometer Algiscan; Drug: Propofol; Drug: Remifentanil
- STANDARD (Sham Comparator): peroperative remifentanil target concentration as standard practice in patients under propofol and remifentanil TCI
  Interventions: Other: Standard practice; Drug: Propofol; Drug: Remifentanil

INTERVENTIONS:
Device: Videopupillometer Algiscan — pupillary diameter measurement every five minutes per-operatively
  Arms: PUPILLO
Other: Standard practice — remifentanil administration left to the discretion of the anesthesiologist in charge according to standard practice
  Arms: STANDARD
Drug: Propofol — TCI
Drug: Remifentanil — TCI

SUMMARY:
The aim of this prospective randomized study was to evaluate the impact of peroperative pupillometry monitoring on per and post-operative opioid consumption in major gynecological surgery. All patients were anesthetized with TCI of propofol and remifentanil. In the intervention group, peroperative remifentanil target was guided by pupillometry. In the other group, remifentanil was administered according to standard practice.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-II
* Elective gynecological surgery
* No ophtalmologic or neurologic disease
* No chronic analgesic medication
* Expected length of surgery 60 minutes minimum

Exclusion Criteria:

* ophtalmologic or neurologic disease
* chronic analgesic medication

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 65 (Actual)
Dates: Start 2010-10; Primary Completion 2012-12 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
peroperative remifentanil consumption in µg/kg/min | duration of surgery

SECONDARY OUTCOMES:
post-operative morphine requirements in mg/kg | 24 hours
  includes initial morphine titration and subsequent PCA use
peroperative propofol consumption in mg/kg/h | duration of surgery

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle Constant, MD-PHD, Study Director — Hôpital Armand Trousseau
Locations (1):
- Departement d'anesthesie Hopital Armand Trousseau, Paris, France